CLINICAL TRIAL: NCT02103517
Title: Risk and Prevention Study: Optimisation of the Preventive Strategies and Evaluation of the Efficacy of n-3 Fatty Acids in Subjects at High Cardiovascular Risk and Suboptimal Health Status
Brief Title: Fish Oil and Cardiovascular Suboptimal Health
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Qiang Zeng, MD, Professor, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2012BAI37B04; N3FACSH (Registry Identifier: n-3 Fatty Acids and Cardiovascular Suboptimal Health)
Record Dates: First submitted 2014-03-27; First posted 2014-04-04 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2017-01

CONDITIONS: Suboptimal Health Status
MeSH Terms: interventions — Docosahexaenoic Acids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Omega-3 fatty acid capsules (Experimental): Omega-3 fatty acid capsules, 4 g/day, requiring intake 2 capsules (1g each one) in the morning and two at night for 3 months.
  Interventions: Dietary Supplement: Omega -3 fatty acids
- corn oil (Placebo Comparator): Corn oil in similar presentation as omega-3 fatty acid capsules, requiring intake 2 capsules in the morning and two at night for 3 months.
  Interventions: Dietary Supplement: Placebo: Corn oil

INTERVENTIONS:
Dietary Supplement: Omega -3 fatty acids — Each subject assigned to active treatment group will receive 4 g/day capsule of omega-3 fatty acids.
  Arms: Omega-3 fatty acid capsules
Dietary Supplement: Placebo: Corn oil — Each subject assigned to the control group will receive 4 g/day capsule of corn oil.
  Arms: corn oil

SUMMARY:
The purpose of this study is to determine whether omega-3 fatty acids supplementation are effective in the improvement of suboptimal health status and cardiovascular risk.

DETAILED DESCRIPTION:
The Suboptimal health status questionnaire (SHSQ-25) is used to evaluate the suboptimal health status. The SHSQ-25 includes 25 questions. The score of the SHSQ-25 is from 0 to 100. Suboptimal health status is defined as the SHSQ-25 score above than 35. The higher scores of the SHSQ-25 one gets, the more severity of suboptimal health status he/she has. All participants are asked to fill in the SHSQ-25 before and after the intervention. If the score decreases after the intervention, it means that the suboptimal health status has been improved.

ELIGIBILITY:
Inclusion Criteria:

1. suboptimal health status, defined as the score of suboptimal health questionnaire ≥35.
2. at least one of cardiovascular risk factors:

   * overweight or obesity, defined as body mass index (BMI) ≥25 kg/m2.
   * systolic blood pressure ≥130 and <140 mmHg and diastolic blood pressure <90 mmHg, or diastolic blood pressure ≥85 and <90 mmHg and systolic blood pressure <140 mmHg
   * fasting plasma glucose ≥100 and <126 mg/dL
   * total cholesterol ≥200 and <240 mg/dL, triglyceride ≥150 and <200 mg/dL, low density lipoprotein-cholesterol ≥130 and <160 mg/dL,and/or high density lipoprotein-cholesterol <40 mg/dL
3. written informed consent

Exclusion Criteria:

1. history of system diseases, such as cardiovascular diseases, digestive system diseases, diseases of respiratory system, blood and immune system diseases, nervous system diseases, endocrine system diseases, and diseases of the genitourinary system.
2. history of mental illness.
3. pregnant or breastfeeding.
4. use of antihypertensive, antidiabetic, or lipid-lowering drugs within the past two weeks.
5. use of fish oil capsules or other supplements containing omega-3 fatty acids within the past two weeks.
6. allergy or intolerance to fish oil, corn oil, omega-3 fatty acids, or vitamin E.
7. participation in another trial.
8. unable to promise to not use drugs and other fish oils during the study.
9. unable to provide informed written consent.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 422 (Actual)
Dates: Start 2014-09; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
the improvement of suboptimal health status | three months
  The improvement of suboptimal health status is evaluated by the change of the SHSQ-25 scores after intervention.
the improvement of traditional cardiovascular risk factors | three months
  To investigate the changes of traditional cardiovascular risk factors such as blood pressure, lipids, fasting plasma glucose, and body mass index with three months supplementation of omega-3 fatty acids. Abnormal cardiovascular risk factors are defined according to the Adult Treatment Panel III criteria for metabolic syndromes and the recommendation by the Working Group on Obesity in China. The number of abnormal cardiovascular risk factors for each participant is recorded before and after intervention. If the number decreases after intervention, it means that the traditional cardiovascular risk factors have been improved.

CONTACTS AND LOCATIONS:
Overall Officials: Qiang Zeng, M.D, Principal Investigator — Chinese PLA General Hospital; Sheng-Yong Dong, M.D, Principal Investigator — Chinese PLA General Hospital
Locations (3):
- China (3):
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - First Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Sichuan Province People's Hospital, Chengdu, Sichuan

REFERENCES:
- [Derived] Zeng Q, Dong SY, Liu YP, Fu J, Shuai P, Zhao ZM, Li TX. Effects of fish oil-derived fatty acids on suboptimal cardiovascular health: A multicenter, randomized, double-blind, placebo-controlled trial. Nutr Metab Cardiovasc Dis. 2017 Nov;27(11):964-970. doi: 10.1016/j.numecd.2017.09.004. Epub 2017 Sep 21. PMID 29066159